CLINICAL TRIAL: NCT07132463
Title: A Multicenter, Randomized Controlled Clinical Study of Concurrent Chemoradiotherapy Followed by Chemotherapy With or Without Tislelizumab for Resectable Ultra-low Rectal Cancer: The RELIEVE-02 Study
Brief Title: Neoadjuvant Chemoradiotherapy Followed by Chemotherapy With or Without Tislelizumab for Resectable Ultra-low Rectal Cancer: The RELIEVE-02 Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELIEVE-02
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer
Keywords: Ultra-low Rectal Cancer; Tislelizumab; Neoadjuvant Chemoradiotherapy; Anus Preservation; PD-1
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent Chemoradiotherapy Followed by Chemotherapy Plus Immunotherapy Group (Experimental): Long-course chemoradiotherapy followed by 4 cycles of CAPOX and Tislelizumab. (Note: Patients evaluated as ncCR after completion, if refusing local excision, may receive an additional 2 cycles of CAPOX and Tislelizumab before re-evaluation.)
  Interventions: Radiation: Long-course chemoradiotherapy; Drug: Tislelizumab combined with the CAPOX regimen
- Concurrent Chemoradiotherapy Followed by Chemotherapy Group (Active Comparator): Long-course chemoradiotherapy followed by 4 cycles of CAPOX. (Note: Patients evaluated as ncCR after completion, if refusing local excision, may receive an additional 2 cycles of CAPOX before re-evaluation.)
  Interventions: Radiation: Long-course chemoradiotherapy; Drug: CAPOX regimen

INTERVENTIONS:
Radiation: Long-course chemoradiotherapy — 45-50.4 Gy in 25-28 fractions to the pelvis on Days 1-5 each week. Capecitabine at a dose of 825 mg/m², taken orally twice daily (bid), 5 days per week during radiotherapy.
Drug: Tislelizumab combined with the CAPOX regimen — Tislelizumab 200 mg IV on Day 1 of each 21-day cycle. Capecitabine: 1000 mg/m² orally twice daily (bid) on Days 1-14 of each 21-day cycle.
  Oxaliplatin: 130 mg/m² IV on Day 1 of each 21-day cycle.
  Arms: Concurrent Chemoradiotherapy Followed by Chemotherapy Plus Immunotherapy Group
Drug: CAPOX regimen — Capecitabine: 1000 mg/m² orally twice daily (bid) on Days 1-14 of each 21-day cycle.
  Oxaliplatin: 130 mg/m² IV on Day 1 of each 21-day cycle.
  Arms: Concurrent Chemoradiotherapy Followed by Chemotherapy Group

SUMMARY:
This open-label, multicenter, randomized controlled trial involved 154 patients with pathologically confirmed, previously untreated, resectable MSI-L or MSS/pMMR ultra-low rectal adenocarcinoma. Patients were randomly assigned (1:1) to two groups to receive concurrent chemoradiotherapy followed by 4-6 cycles of chemotherapy ± tislelizumab. After treatment, patients who achieved complete clinical response (cCR), including those who reached pCR after local excision, or near cCR with pCR after local excision, were recommended to continue with 4-2 cycles of chemotherapy ± tislelizumab, followed by a watch-and-wait approach. Patients evaluated as incomplete responders were recommended for total mesorectal excision (TME) surgery. The primary endpoint is the anus preservation rate, while secondary endpoints include CR rate, 1-year/2-year/3-year organ preservation rates, 1-year/2-year/3-year EFS rates, and 1-year/2-year/3-year OS rates, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent, understand, and comply with the requirements and evaluation schedule.
2. Age ≥18 and ≤75 years old.
3. Histologically confirmed rectal adenocarcinoma.
4. Immunohistochemistry confirmed pMMR (positive for MLH1, MSH2, MSH6, and PMS2), or PCR/NGS confirmed MSI-L or MSS.
5. Tumor distal margin confirmed to be ≤ 3 cm from the anal verge by colonoscopy, digital rectal examination, or MRI.
6. Clinical stage cT1-3N1M0 or cT3N0M0 (the 8th UICC/AJCC; T and N evaluated by MRI).
7. Resectable primary tumor assessed by the Investigator.
8. No prior anti-tumor treatment for rectal cancer.
9. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
10. Adequate organ function.
11. Female subjects with the ability to become pregnant must have a serum pregnancy test with a negative result within 72 hours before the first dose and be willing to use highly effective contraceptive methods during the trial and for 120 days after the last dose. Male subjects whose partners are women of childbearing potential should be surgically sterilized or agree to use a highly effective method of contraception during the trial and for 120 days after the last dose.

Exclusion Criteria:

1. Histologically confirmed poorly differentiated/undifferentiated adenocarcinoma, mucinous adenocarcinoma, or signet ring cell carcinoma.
2. Previously received treatment for rectal cancer or have evidence of distant metastasis.
3. Presence of the following high-risk factors assessed by MRI: MRF+, EMVI+, cN2, positive lateral lymph nodes, T3d.
4. Presence of or at high risk for obstruction, perforation, or bleeding.
5. Unsuitability for long-course radiotherapy.
6. Inability to tolerate surgery.
7. ≥ 2 colorectal cancer lesions at the same time.
8. Contraindications for MRI examination.
9. Other malignant tumors in the past or currently present.
10. Active autoimmune disease requiring systemic therapy within the past 2 years.
11. HIV infection.
12. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers (HBV DNA > 500 IU/mL) or active HCV carriers with detectable HCV RNA.
13. Hypersensitivity to any ingredient of tislelizumab, capecitabine, and oxaliplatin, or to any component of their containers.
14. Other conditions judged by the researcher as not meeting the enrollment requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 154 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Anus preservation rate | From first dose of radiotherapy up to approximately 24/32±4 weeks.
  Defined as the anus preservation rate in the efficacy-evaluable analysis set of patients, as assessed by the investigators.

SECONDARY OUTCOMES:
Complete Response rate (CR Rate) | From first dose of radiotherapy up to approximately 24/32±4 weeks.
  Defined as the proportion of participants with clinical complete response (cCR) and pathologic complete response (pCR), determined by the investigators.
1/2/3-Year Organ-Preservation Rate | From first dose of radiotherapy up to approximately 36 months.
  Defined as the proportion of participants who survived and did not undergo TME at 1, 2, and 3 years.
1/2/3-Year EFS Rate | From first dose of radiotherapy up to approximately 36 months.
  Defined as the proportion of participants who did not develop local recurrence, distant metastasis, new invasive primary lesions of colorectal cancer, or death at 1, 2, and 3 years.
1/2/3-Year OS Rate | From first dose of radiotherapy up to approximately 36 months.
  Defined as the proportion of participants who survived at 1, 2, and 3 years.
Percentage of Participants With Adverse Events | From first dose of radiotherapy up to approximately 36 months.
  Percentage of participants with adverse events (AEs), immune-related adverse events(irAE), and serious adverse events (SAEs).